CLINICAL TRIAL: NCT01628276
Title: Brain Functional Connectivity Changes Following Cognitive Rehabilitation in Multiple Sclerosis: an fMRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sina Hospital, Iran (Other)
Responsible Party: Principal Investigator, Mohammad Ali Sahraian, Vice President, Sina Hospital, Iran
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MSRC-AE-DCM-1
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: MS (Multiple Sclerosis)
Keywords: Multiple Sclerosis; MRI Scans
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rehab first (Experimental)
  Interventions: Behavioral: Cog Rehab
- Rehab Second (Experimental)
  Interventions: Behavioral: Cog Rehab
- Non Rehab (No Intervention)

INTERVENTIONS:
Behavioral: Cog Rehab — Cognitive rehab for MS patients
  Arms: Rehab Second; Rehab first

SUMMARY:
This trial seeks to investigate brain network changes following cognitive rehabilitation in MS patients. The investigators hypothesize that rehabilitation interventions improve connectivity in the brain.Novel Magnetic Resonance Imaging technique is performed to investigate changes in brain plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Definitive MS diagnosis
* Right handedness
* EDSS 0-4
* No relapse in past 6 weeks
* Willing to consent and participate in the study

Exclusion Criteria:

* Pregnancy
* Left handedness
* Neurologic or psychiatric disorder other than MS

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
functional connectivity | 0, 2nd, 4th Month
  Changes in correlation of brain activity in different regions of brain as assessed by Blood Oxygenation Level Dependent (BOLD) signal

CONTACTS AND LOCATIONS:
Locations (1):
- Sina Hospital, Tehran, Tehran Province, Iran